CLINICAL TRIAL: NCT02852772
Title: Does Micro-albuminuria is a Predictive Factor for Cognitive Impairment in Persons Living With HIV (PLHIV) Who Achieve cART-sustained Immunovirological Control ?
Acronym: ALCOVE
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: AMR_2014-2
Record Dates: First submitted 2016-07-26; First posted 2016-08-02 (Estimated); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: HIV
Keywords: Cognitive impairment; HIV; Microalbuminuria; Chronic kidney disease
MeSH Terms: conditions — Cognitive Dysfunction; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- PLHIV with microalbuminuria: Patient infected with HIV and well controlled by treatments, with microalbuminuria for at least 5 years
  Interventions: Behavioral: Cognitive function tests
- PLHIV without microalbuminuria (control): Patient infected with HIV and well controlled by treatments, without microalbuminuria, matched for age +/- 5 years
  Interventions: Behavioral: Cognitive function tests

INTERVENTIONS:
Behavioral: Cognitive function tests

SUMMARY:
Chronic kidney disease (CKD), frequent in PLHIV, is a risk factor for cognitive impairment. Micro-albuminuria is an early manifestation of CKD and a marker of vascular risk, notably affecting the small vessels. In the older general population microalbuminuria is associated with greater annual cognitive decline and has been proposed as an easily and inexpensive measured marker predicting future cognitive function decline. Ageing of the PLH leads to an increase of cognitive disorders and chronic renal failure incidence and could imply a common underlying mechanism affecting the renal and cerebral microvasculature. In this setting the investigators undertake this prospective, cross-sectional, case-control study to determine whether the presence of a microalbuminuria at least 5 years ago in PLHs with sustained good combination antiretroviral therapy (cART)-controlled immunovirological parameters could be a marker predicting future cognitive impairment. They chose PLHs infected for at least 5 years and with cART-sustained immunovirological control for at least 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Known HIV infection for at least 5 years
* Undetectable viral load under antiretroviral (ARV) treatment for at least 1 year, regardless of the type of ARV
* Number of CD4 ≥ 350, regardless of the CD4 nadir
* Unopposed to participate to the study

For cases

- Micro-albuminuria defined by microalbuminuria / creatinuria between 3 and 30 mg/mmol

For controls, matched for age +/- 5 years - Absence of microalbuminuria defined by microalbuminuria / creatinuria <3 mg/mmol

Exclusion criteria

* Known neurological disease, active or former
* Active and regular use of drugs
* Active Chronic alcoholism
* Diabetes with known complications
* Renal failure with glomerular filtration rate <15 ml / min
* Micro-albuminuria / creatinuria> 30 mg / mmol
* HIVAN
* Unbalanced arterial hypertension
* Patient did not have dosing glucose and lipid levels in over a year
* Unaffiliated patient (or copyright holder) to a social security scheme
* People enjoying a measure of legal protection Pregnant or breastfeeding

Secondary exclusion criteria

- Neurological disease found during the assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients registered in the HIVREINE database (which combines nephrology and infectious diseases services of AP-HP, Greater Paris University Hospitals)
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2014-07; Primary Completion 2016-11-07 (Actual); Study Completion 2016-11-07 (Actual)

PRIMARY OUTCOMES:
Z-Score of five neurocognitive domains tested and global deficit score | 4 hours
  Comparisons of composite cognitive scores (z-score) and scores of global cognitive deficits (GDS) between the two populations. The neuropsychological tests are made during a single consultation of a half day.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation Ophtalmologique Adolphe de Rothschild, Paris, France